CLINICAL TRIAL: NCT06456008
Title: Prospective Registry of Outcome and Correlates of Chemosensory Dysfunction at the Smell & Taste Clinic of UZ Leuven
Brief Title: Prospective Registery of Smell/Taste Clinic Ear/Nose/Throat
Acronym: ProspeRo'Scent
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S67158
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Olfactory Disorder; Taste Disorders; Smell Dysfunction; Smell Disorder
MeSH Terms: conditions — Taste Disorders; Olfaction Disorders | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard of care — Standard of care

SUMMARY:
Smell/taste disorders are common conditions with a significant impact on quality of life. In September 2021, a specific consultation for patients with smell and taste disorders was initiated at the ENT-HNS (ear, nose, and throat, head and neck surgery) department of UZ Leuven, partly in light of post-COVID-19 related smell disorders.

With this observational ambidirectional study, the investigators aim to better map smell/taste disorders in the Belgian/Flemish population. Using standard-of-care diagnostic tests and structured questionnaires, the investigators strive to gain more insight into the severity, impact, and progression/prognosis of smell/taste disorders.

ELIGIBILITY:
Inclusion criteria:

* The psychophysical testing as well as the questionnaires require a cooperative participant who can understand and follow instructions and communicate their choices.
* Informed consent is necessary upon participation for prospective registry.

There are no exclusion criteria related to sex, gender, or ethnicity. There are no exclusion criteria related to medical history or prior treatments.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients consulting for chemosensory dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Chemosensory function | Observational up to 5 years follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- UZ/KU Leuven, Leuven, Vlaams-Brabant, Belgium